CLINICAL TRIAL: NCT06943872
Title: A Phase 3 Randomized, Open-Label, Multicenter Study of Sonrotoclax Plus Anti-CD20 Antibody Therapies Versus Venetoclax Plus Rituximab in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: A Study to Investigate Progression-Free Survival With Sonrotoclax Plus Obinutuzumab Or Sonrotoclax Plus Rituximab Compared With Venetoclax Plus Rituximab Treatment In Patients With Relapsed and/or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CELESTIAL-RRCLL)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Collaborators: German CLL Study Group (Other)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-11417-303; 2024-517131-52-00 (EU CTIS Number); CLL-RR1 (Other: German CLL Study Group)
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: B-cell lymphoma 2 inhibitor (BCL-2i); CLL-RR1; German CLL Study Group
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab; Rituximab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Sonrotoclax plus Obinutuzumab (Experimental): Sonrotoclax and obinutuzumab will be administered in combination.
  Interventions: Drug: Sonrotoclax; Drug: Obinutuzumab
- Arm B: Sonrotoclax plus Rituximab (Experimental): Sonrotoclax and rituximab will be administered in combination.
  Interventions: Drug: Sonrotoclax; Drug: Rituximab
- Arm C: Sonrotoclax plus Obinutuzumab (MRD) (Experimental): Sonrotoclax and obinutuzumab will be administered in combination with treatment guided by evaluation of minimal residual disease (MRD).
  Interventions: Drug: Sonrotoclax; Drug: Obinutuzumab
- Arm D: Venetoclax plus Rituximab (Active Comparator): Venetoclax and rituximab will be administered in combination.
  Interventions: Drug: Rituximab; Drug: Venetoclax

INTERVENTIONS:
Drug: Sonrotoclax — Administered orally
  Other Names: BGB-11417
  Arms: Arm A: Sonrotoclax plus Obinutuzumab; Arm B: Sonrotoclax plus Rituximab; Arm C: Sonrotoclax plus Obinutuzumab (MRD)
Drug: Obinutuzumab — Administered intravenously
  Other Names: Gazyva
  Arms: Arm A: Sonrotoclax plus Obinutuzumab; Arm C: Sonrotoclax plus Obinutuzumab (MRD)
Drug: Rituximab — Administered intravenously
  Other Names: Rituxan
  Arms: Arm B: Sonrotoclax plus Rituximab; Arm D: Venetoclax plus Rituximab
Drug: Venetoclax — Administered Orally
  Other Names: Venclexta
  Arms: Arm D: Venetoclax plus Rituximab

SUMMARY:
The goal of this study is to compare how well sonrotoclax plus obinutuzumab works versus venetoclax plus rituximab in treating adults with relapsed and/or refractory (R/R) chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL). The study will also compare how well sonrotoclax plus rituximab works versus venetoclax plus rituxumab in treating adults with R/R CLL/SLL. The safety of these treatments will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CLL/SLL that meets the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria
* Received one or more prior therapies for CLL/SLL. For each line of therapy, participants must have received at least 2 cycles of the therapy
* Participants with prior BCL2i exposure are eligible if remission duration was ≥3 years with ≥2 years from last BCL2i intake
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1, or 2
* Adequate organ function

Exclusion Criteria:

* Known active prolymphocytic leukemia or currently suspected Richter's transformation
* Prior autologous stem cell transplantation or chimeric antigen receptor T-cell therapy within 3 months before first dose of study drug
* Prior allogeneic stem cell transplant with active graft-versus-host disease (GVHD), requiring immunosuppressive drugs for treatment of GVHD, or have taken calcineurin inhibitors within 4 weeks prior to consent
* Known central nervous system involvement by CLL/SLL
* Severe or debilitating pulmonary disease
* Clinically significant cardiovascular disease

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) as assessed by Blinded Independent Review Committee (BIRC) for Arm A versus Arm D | Up to approximately 51 months
  PFS is defined as the time from randomization to the date of progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) as assessed by BIRC for Arm B versus Arm D | Up to approximately 69 months
  PFS is defined as the time from randomization to the date of progression or death, whichever occurs first.
Rate of uMRD4 for Arm A versus Arm D | Up to approximately 12 months
  The rate of undetectable minimal residual disease (uMRD4) in peripheral blood based on next-generation sequencing (NGS)
Complete Response Rate as assessed by BIRC for Arm A versus Arm D | Up to approximately 25 months
  Complete Response Rate (CRR) is defined as the percentage of participants that achieve a best response of complete response (CR) or complete response with incomplete hematopoietic recovery (CRi)
Overall Survival for Arm A versus Arm D | Up to approximately 84 months
  Overall survival (OS) is defined as the time from the date of randomization to the date of death
PFS per Investigator Assessment (INV) for Arm B versus Arm D | Up to approximately 69 months
  PFS is defined as the time from randomization to the date of progression or death, whichever occurs first.
CRR per BIRC and by INV for Arm B versus Arm D | Up to approximately 25 months
  CRR is defined as the percentage of participants that achieve a best response of CR or CRi
OS for Arm B versus Arm D | Up to approximately 84 months
  OS is defined as the time from the date of randomization to the date of death
Rate of uMRD4 for Arm B versus Arm D | Up to approximately 25 months
  The rate of uMRD4 in peripheral blood based on NGS
PFS per BIRC and by INV for Arm A versus Arm B | Up to approximately 69 months
  PFS is defined as the time from randomization to the date of progression or death, whichever occurs first.
CRR per BIRC and by INV for Arm A versus Arm B | Up to approximately 25 months
  CRR is defined as the percentage of participants that achieve a best response of CR or CRi
OS for Arm A versus Arm B | Up to approximately 84 months
  OS is defined as the time from the date of randomization to the date of death
Rate of uMRD4 for Arm A versus Arm B | Up to approximately 25 months
  The rate of uMRD4 in peripheral blood based on NGS
Rate of uMRD4 for Arm A versus Arm D | Up to approximately 25 months
  The rate of uMRD4 in peripheral blood based on NGS
CRR per INV for Arm A versus Arm D | Up to approximately 25 months
  CRR is defined as the percentage of participants that achieve a best response of CR or CRi
PFS per INV for Arm A versus Arm D | Up to approximately 51 months
  PFS is defined as the time from randomization to the date of progression or death, whichever occurs first.
PFS per INV for Arm C versus Arm D | Up to approximately 69 months
  PFS is defined as the time from randomization to the date of progression or death, whichever occurs first.
CRR per INV for Arm C versus Arm D | Up to approximately 25 months
  CRR is defined as the percentage of participants that achieve a best response of CR or CRi
OS for Arm C versus Arm D | Up to approximately 84 months
  OS is defined as the time from the date of randomization to the date of death
Rate of uMRD4 for Arm C versus Arm D | Up to approximately 25 months
  The rate of uMRD4 in peripheral blood based on NGS
Overall Response Rate (ORR) per BIRC and by INV | Up to approximately 25 months
  ORR is defined as the percentage of participants that achieve a best response of partial response (PR) or better
Duration of Response (DOR) per BIRC and by INV | Up to approximately 69 months
  DOR is defined as the time from the date that response criteria were first met to the date of first documentation of disease progression or death, whichever occurs first
Time to Response (TTR) per BIRC and by INV | Up to approximately 25 months
  TTR is defined as the time from the date of randomization to the date response criteria were first met
Time to Next Anti-CLL/SLL Treatment (TTNT) | Up to approximately 84 months
  TTNT is defined as the time from the date of randomization to the date of next anti-CLL/SLL treatment
Rate of uMRD4 | Up to approximately 25 months
  The rate of uMRD4 in peripheral blood based on NGS
Change from Baseline in the European Organisation of Research and Treatment of Cancer-Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30) Global Health Status/Quality of Life and Physical Functioning Scales | Baseline and up to approximately 69 months
  The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 =Not at all (best) to 4 =Very Much (worst) and 2 questions answered on a 7-point scale where 1 =Very poor (worst) to 7 =Excellent (best). Higher scores in global health status (GHS) and functional scales indicate better health-related quality of life (HRQoL).
Change from Baseline in EORTC QLQ for Chronic Lymphocytic Leukemia (EORTC QLQ-CLL17) Symptom Burden and Fatigue Scales | Baseline and up to approximately 69 months
  The EORTC QLQ-CLL17 is the CLL module of QLQ-C30 consisting of 17 items and comprising 3 scales: symptom burden due to disease and/or treatment (6 items), physical condition/fatigue (4 items), and worries/fears about health and functioning (7 items) Items are rated using a 4-point response scale ("not at all," "a little," "quite a bit," and "very much") and the recall period for all items is the past 7 days. Lower scores indicate better HRQoL.
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | From the first dose of study drug(s) to 30 days after the last dose of sonrotoclax or venetoclax, or 90 days after the last dose of obinutuzumab or rituximab; up to approximately 26 months
  Number of participants with TEAEs, including laboratory values, vital signs, and physical examination findings, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (108):
- United States (26):
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute, Palo Alto, California
  - Scripps Prebys Cancer Center, San Diego, California
  - Rocky Mountain Cancer Centers (Williams) Usor, Aurora, Colorado
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology, Norwich, Connecticut
  - Northwestern University, Chicago, Illinois
  - Illinois Cancer Specialists (Niles) Usor, Niles, Illinois
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - The Cancer and Hematology Centers, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center Mskcc, New York, New York
  - Clinical Research Alliance, Inc, Westbury, New York
  - University of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Levine Cancer Center, Charlotte, North Carolina
  - Oncology Hematology Care Clinical Trials, Llc, Cincinnati, Ohio
  - Oncology Associates of Oregon Willamette Valley Cancer Center, Eugene, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Upmc Hillman Cancer Center(Univ of Pittsburgh), Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology Baylorcharles A Sammons Cancer Center, Dallas, Texas
  - Texas Oncology San Antonio Medical Center Usor, San Antonio, Texas
  - Texas Oncology Tyler, Tyler, Texas
  - Northwest Cancer Specialist, Pc(Us Oncology Research), Vancouver, Washington
- Australia (13):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Northern Nsw Health District, Lismore, New South Wales
  - Macquarie University, North Ryde, New South Wales
  - Genesiscare North Shore, St Leonards, New South Wales
  - Sunshine Coast Hospital and Health Service, Birtinya, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Health, Clayton, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Rockingham Hospital, Cooloongup, Western Australia
  - Perth Blood Institute, West Perth, Western Australia
- Hanusch Krankenhaus, Vienna, Austria
- Brazil (14):
  - CETUS, Belo Horizonte
  - Universidade de Campinas Centro de Hematologia E Hemoterapia, Campinas
  - Hospital Erasto Gaertner, Curitiba
  - Complexo Hospitalar de Niteroi, Niterói
  - Irmandade Da Santa Casa de Misericordia Hospital Porto Alegre, Porto Alegre
  - Hospital Sao Lucas, Rio de Janeiro
  - Instituto Dor de Pesquisa E Ensino Rio de Janeiro, Rio de Janeiro
  - Hospital Santa Izabel, Salvador
  - Hospital Samaritano Sao Paulo, São Paulo
  - Hospital Nove de Julho Dasa, São Paulo
  - Instituto Brasileiro de Controle Do Cancer, São Paulo
  - Instituto Dor de Pesquisa E Ensino Sao Paulo, São Paulo
  - Hcfmusp Servico de Hematologia, Hemoterapia E Terapia Celular, São Paulo
  - Hospital Santa Rita de Cassia Afecc, Vitória
- China (13):
  - China Japan Friendship Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospitalqishan Branch, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Guangzhou First Peoples Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital Wuxiang Branch, Nanning, Guangxi
  - Affiliated Hospital of Jiangnan University South Campus, Wuxi, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Shaanxi Provincial Peoples Hospital, Xi'an, Shaanxi
  - Jining No Peoples Hospital West Branch, Jining, Shandong
  - The Affiliated Hospital of Qingdao University Branch West Coast, Qingdao, Shandong
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
- Czechia (2):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense C
- France (6):
  - Chu Clermont Ferrand Therapie Cellulaire and Hematolo, Clermontferrand
  - Centre Hospitalier Universitaire Nantes Hotel Dieu, Nantes
  - Hopital de La Pitie Salpetriere, Paris
  - Hopital Robert Debre, Reims
  - Chu Rennes, Rennes Cedes
  - Centre Henri Becquerel, Rouen
- Germany (6):
  - Osp Kurfuerstendamm, Berlin
  - Uniklinik Koeln (Aoer), Cologne
  - Universitatsklinikum Jena Klinik Fur Innere Medizin Ii, Jena
  - Stauferklinikum Schwabisch Gmund Kliniken Ostalb, Mutlangen
  - Dietrich Bonhoeffer Klinikum Neubrandenburg, Neubrandenburg
  - Haematologisch Onkologische Schwerpunktpraxis, Würzburg
- St Jamess Hospital, Dublin, Ireland
- Italy (2):
  - Ao Brotzu Ospedale Oncologico Armando Businco, Cagliari
  - Ospedale San Raffaele, Milan
- Albert Schweitzer Ziekenhuis, Dordrecht, Netherlands
- New Zealand (2):
  - North Shore Hospital, Auckland
  - Auckland City Hospital, Auckland
- South Korea (7):
  - Pusan National University Hospital, Seogu, Busan Gwang'yeogsi
  - Seoul National University Bundang Hospital, BundangGu SeongnamSi, Gyeonggi-do
  - National Cancer Center (Korea), IlsandongGu GoyangSi, Gyeonggi-do
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St Marys Hospital, SeochoGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
- Spain (7):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de La Princesa, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Costa Del Sol (Marbella, Malaga), Marbella
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Virgen de Valme (Sevilla), Seville
- United Kingdom (5):
  - University Hospitals Dorset Royal Bournemouth Hospital, Bournemouth
  - Kings College Hospital, London
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Freeman Hospital, Newcastle upon Tyne
  - Royal Cornwall Hospitalsnhs Trust, Truro

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/